CLINICAL TRIAL: NCT01310257
Title: Evaluation of Questionnaire Measures for Patients With Osteoarthritis of the Knee
Brief Title: Measures of Pain Relevant to Knee Osteoarthritis
Status: Completed | Type: Observational
Sponsor: University of Nottingham (Other)
Collaborators: Arthritis Research UK (Other)
Responsible Party: Sponsor
Other Study IDs: 10052; 9227 (Registry Identifier: UKCRN)
Record Dates: First submitted 2011-03-02; First posted 2011-03-08 (Estimated); Last update posted 2014-01-17 (Estimated); Status verified 2014-01

CONDITIONS: Osteoarthritis of the Knee
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Knee osteoarthritis: Patients will have osteoarthritis (OA) of the knee defined and scored radiologically in Study 1. Patients in Study 2 will also have OA of the knee, but a clinical diagnosis will suffice. All patients will report knee pain.
  Interventions: Other: Questionnaires

INTERVENTIONS:
Other: Questionnaires — Patients will be given questionnaires relevant to their condition to complete. In Study 2 and a sub-study of Study 1, patients will be invited to take part in Quantitative Sensory Testing.

SUMMARY:
The aim is to improve understanding of the assessment of pain experience in patients with osteoarthritis (OA) of the knee. The current study will be divided into two parts. In Study 1, the investigators will analyse existing questionnaires relevant to the mechanisms and therapeutic targets of knee OA to establish discrete dimensions that discriminate between the different mechanisms of pain. On the basis of this analysis, the investigators will refine the questionnaires to maximise their sensitivity to knee OA. In Study 2, the investigators will seek to confirm the factor structure identified in the questionnaires in Study 1 and explore potential mediator and moderator variables between pain and quality of life using the refined measures. The investigators will also evaluate Quantitative Sensory Testing as a predictor of OA knee pain.

ELIGIBILITY:
Inclusion Criteria:

* Participants in Study 1 will have OA of the knee defined and scored radiologically and will report knee pain. Participants in Study 2 will also have OA of the knee, but a clinical diagnosis will suffice.

Exclusion Criteria:

* Inability to speak or understand English
* Under the age of 18 years old
* knee joint surgery within three months prior to participation
* Diagnosed Rheumatoid Arthritis, Psoriatic Arthritis, Gout or any other inflammatory arthritis disorder
* The participants in Study 2 will also be excluded if they participated in Study 1

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We aim to recruit a cross section of participants covering a broad spectrum of people with OA of the knee. Community participants will be identified from a cohort of patients who have already agreed to be contacted about future research studies. Additional participants will be identified from clinics at Nottingham University Hospitals and Sherwood Forest Hospitals NHS Foundation Trust, GP surgeries in the local area and patients on a knee OA pathway from Nottingham Healthcare partnership. These sources of recruitment will include those attended rheumatology and orthopaedic specialist clinics for knee OA and rheumatology outpatients at the Queens Medical Centre (QMC)
Sampling Method: Non-Probability Sample
Enrollment: 448 (Actual)
Dates: Start 2010-12; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Questionnaire set assessing physical symptoms, cognitive and emotional factors, and quality of life in knee OA. | Patients will be assessed after diagnosis of OA of the knee. There is no specific time point after diagnosis, because we are interested in a broad spectrum of patients with OA of the knee. All patients will be assessed at enrollment into the study.
  Patients will be given a questionnaire set assessing pain (nociceptive and neuropathic), anxiety, depression, fatigue, illness belief, pain self-efficacy, coping, helplessness and quality of life, associated with OA of the knee. The psychometric properties of the questionnaire set will be reported, including results from Rasch Analysis, Cronbach's Alpha and results from Factor Analysis.

SECONDARY OUTCOMES:
Quantitative Sensory Testing assessing pain and sensory thresholds for a noxious stimulus (Pain Pressure Thresholds) | Patients will be assessed after diagnosis of OA of the knee. There is no specific time point after diagnosis, because we are interested in a broad spectrum of patients with OA of the knee.
  Pain and sensory thresholds will be reported for the affected area (i.e., OA knee) and control areas (e.g., healthy contralateral knee).

CONTACTS AND LOCATIONS:
Overall Officials: Bryan Moreton, Principal Investigator — University of Nottingham
Locations (3):
- United Kingdom (3):
  - Nottingham Country Health Partnerships, Nottingham
  - Nottingham University Hospitals NHS Trust, Nottingham
  - Sherwood Forest Hospitals NHS Trust, Nottingham

REFERENCES:
- See also: Arthritis Research UK Pain Centre — http://www.nottingham.ac.uk/paincentre/index.aspx